CLINICAL TRIAL: NCT07181694
Title: A Double-Blind, Comparative, Randomized Clinical Study of the Pharmacokinetics, Safety, and Immunogenicity of Single Subcutaneous Doses of BCD 057 100 mg/mL, BCD-057 50 mg/mL, and Humira 100 mg/mL in Healthy Subjects
Brief Title: A Study of Pharmacokinetics, Safety, and Immunogenicity of BCD-057 100 mg/mL, BCD-057 50 mg/mL, and Humira 100 mg/mL in Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: BCD-057-5
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Healthy Adult Male
Keywords: Tumor Necrosis Factor Inhibitors; Anti-Inflammatory Agents; Adalimumab; Monoclonal Antibody; Pharmacokinetics
MeSH Terms: interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ADA100 (Experimental): Subjects will receive a single subcutaneous injection of BCD-057 at a dose of 40 mg/0.4 mL
  Interventions: Drug: Adalimumab (BCD-057) 100 mg/mL
- ADA50 (Active Comparator): Subjects will receive a single subcutaneous injection of BCD-057 at a dose of 40 mg/0.8 mL
  Interventions: Drug: Adalimumab (BCD-057) 50 mg/mL
- HUM100 (Active Comparator): Subjects will receive a single subcutaneous injection of Humira at a dose of 40 mg/0.4 mL
  Interventions: Drug: Adalimumab (Humira) 100 mg/mL

INTERVENTIONS:
Drug: Adalimumab (BCD-057) 100 mg/mL — Single subcutaneous injection
  Arms: ADA100
Drug: Adalimumab (BCD-057) 50 mg/mL — Single subcutaneous injection
  Arms: ADA50
Drug: Adalimumab (Humira) 100 mg/mL — Single subcutaneous injection
  Arms: HUM100

SUMMARY:
The aim of this study is to establish comparability of pharmacokinetic parameters and similarity of the safety and immunogenicity profiles of single subcutaneous doses of BCD 057 100 mg/mL and BCD-057 50 mg/mL, as well as BCD-057 100 mg/mL and Humira 100 mg/mL, in healthy subjects. The study is conducted in a population of healthy male subjects aged 18-45 years inclusive at the time of signing the ICF, with a body mass index in the range of 18.5 to 30.0 kg/m2.

DETAILED DESCRIPTION:
The study includes following periods:

* Screening (not more than 14 days)
* Main period (Day 1 to Day 71)

Subjects meeting the eligibility criteria will be randomized with equal probability into one of three groups:

* ADA100 group - subjects will receive a single subcutaneous injection of BCD-057 at a dose of 40 mg/0.4 mL
* ADA50 group - subjects will receive a single subcutaneous injection of BCD-057 at a dose of 40 mg/0.8 mL
* HUM100 group - subjects will receive a single subcutaneous injection of Humira at a dose of 40 mg/0.4 mL

During randomization, subjects will be stratified by the following criterion:

* Body weight (<75 kg or ≥75 kg)

ELIGIBILITY:
Inclusion Criteria:

1. Signing the Informed Consent Form of the study.
2. Men aged 18-45 years inclusive at the time of signing the Informed Consent Form.
3. Body mass index (BMI) in the range of 18.5-30.0 kg/m2.
4. The confirmed "healthy" status based on the conventional clinical and laboratory assessments and investigations obtained as screening.
5. Hemodynamic parameters within the normal range: systolic blood pressure (SBP) in the range of 100-130 mmHg, diastolic (DBP) in the range of 60-90 mmHg, wrist pulse rate 60-90 bpm, obtained at screening.
6. ECG data normal for the age (no ischemia, arrhythmia, conduction disorders).
7. No chronic infections (HIV, hepatitis B or C) and no history of chronic inflammatory diseases.
8. No signs of active or latent tuberculosis according to screening X-ray and tuberculosis test results.
9. No acute infections within 4 weeks prior to the date of randomization.
10. The ability of the subject to follow the Protocol procedures, according to the Investigator.
11. No history of alcoholism or drug addiction and negative test results for alcohol, psychotropic and narcotic substances, psychoactive drugs at screening and before the IP administration.
12. Willingness of subjects to use condoms during any sexual contact by penetration with persons of any sex, including pregnant women, starting from the signing of the Informed Consent Form, during the study and for 5 months after the IP administration. This requirement does not apply to subjects who have undergone surgical sterilization (bilateral orchiectomy).
13. Willingness to refuse to donate sperm and conceive a child starting from the signing of the Informed Consent Form, during the study and for 5 months after the IP administration.
14. Willingness not to drink alcohol within 24 hours before and after the IP administration, within 24 hours before each scheduled visit.
15. Willingness to refrain from smoking within 2 hours before the IP administration and then 2 hours before each measurement of blood pressure (BP), wrist pulse rate, respiratory rate, blood sampling, ECG.
16. Willingness to refrain from vaccination with live attenuated vaccines (e.g., intranasal influenza, measles, mumps, rubella, polio, BCG, yellow fever, chickenpox, and typhoid TY21a vaccines) throughout the study.
17. Willingness to refrain from taking any medications, including over-the-counter drugs, vitamins and food supplements, with the exception of drugs prescribed by the Investigator for the treatment of AEs, throughout the study.

Exclusion Criteria:

1. Mental illness or other conditions that may, in the Investigator's opinion, affect the subject's ability to comply with the Study Protocol.
2. Any significant, in the Investigator's opinion, surgical procedures performed less than 30 days before the screening examination and potentially affecting clinical study results.
3. A history of allergic reactions (anaphylactic shock or multiple drug allergy according to the Investigator's assessment).
4. Known allergy or intolerance to monoclonal antibody products (murine, chimeric, humanized, fully human) or any other components of the IP.
5. Impossibility of installing a venous catheter for collecting blood samples (e.g., due to skin disorders at the venipuncture sites).
6. Administration and use of the following drugs:

   1. Past use of adalimumab or any other drugs that inhibit tumor necrosis factor alpha.
   2. Regular oral or parenteral administration of any medicinal products, including over-the-counter drugs, vitamins, and dietary supplements, less than 14 days prior to the estimated date of randomization.
   3. Taking medications, including over-the-counter drugs, which have a pronounced effect on hemodynamics and liver function (barbiturates, omeprazole, cimetidine, etc.), less than 30 days before the estimated date of randomization.
   4. Using drugs that affect the immune status (cytokines and their inducers, glucocorticoids, etc.) less than 30 days before the estimated date of randomization.
   5. Systemic use of antibacterial, antifungal, antiviral or antiprotozoal drugs less than 30 days before the estimated date of randomization.
   6. Vaccination with live attenuated vaccines within 4 weeks before the estimated date of randomization.
7. Positive results of screening tests for HIV, hepatitis B and C viruses.
8. Results of conventional laboratory tests or investigations out of the reference ranges accepted at the study sites.
9. Chronic diseases of the cardiovascular, bronchopulmonary, neuroendocrine systems, as well as diseases of the gastrointestinal tract, kidneys, blood.
10. Acute infectious diseases less than 4 weeks before the estimated date of randomization, as well as chronic and other diseases that, in the Investigator's opinion, may affect the pharmacokinetics, safety, and immunogenicity of the IP.
11. Smoking more than 10 cigarettes a day.
12. Consumption of more than 10 units of alcohol per week (1 unit of alcohol is equivalent to ½ L of beer, 200 mL of wine or 50 mL of spirits) or a history of alcoholism, drug addiction, or drug abuse.of blood or plasma within 60 calendar days prior to the expected date of randomization.
13. Donation of ≥450 mL of blood or plasma within 60 calendar days prior to the expected date of randomization.
14. Participation in any clinical studies in less than 90 calendar days before the date of randomization, if the subject received a medicinal product during the clinical study.
15. Previous participation in the same study if the subject was randomized and received the IP during the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 444 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
AUC(0-∞) | Before drug administration and 1, 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 336, 672, 1008, 1440, 1680 hours after drug administration
  Area Under the Plasma Concentration-time Curve From Zero (0) to Time Infinity
Cmax | Before drug administration and 1, 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 336, 672, 1008, 1440, 1680 hours after drug administration
  Maximum Concentration

SECONDARY OUTCOMES:
AUC(0-1680) | Before drug administration and 1, 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 336, 672, 1008, 1440, 1680 hours after drug administration
  Area Under the Plasma Concentration-time Curve From Zero (0) Hours to 1680 Hours
Tmax | Before drug administration and 1, 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 336, 672, 1008, 1440, 1680 hours after drug administration
  Time to Reach Maximum Concentration
T½ | Before drug administration and 1, 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 336, 672, 1008, 1440, 1680 hours after drug administration
  Half-life Period
Vd | Before drug administration and 1, 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 336, 672, 1008, 1440, 1680 hours after drug administration
  Volume of Distribution
Kel | Before drug administration and 1, 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 336, 672, 1008, 1440, 1680 hours after drug administration
  Elimination Rate Constant
Cl | Before drug administration and 1, 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 336, 672, 1008, 1440, 1680 hours after drug administration
  Clearance

CONTACTS AND LOCATIONS:
Overall Officials: Arina V Zinkina-Orikhan, Study Director — Biocad
Locations (3):
- Russia (3):
  - I.M. Sechenov First Moscow State Medical University, Moscow
  - LLC "X7 Clinical Research", Saint Petersburg
  - LLC "Research Center Eco-Safety", Saint Petersburg